CLINICAL TRIAL: NCT07140978
Title: A Clinical Trial to Evaluate the Efficacy of a Healthy Meal Plan in Improving Health Biomarkers and Promoting Healthy Weight Management.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Green Chef Corporation (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20678
Record Dates: First submitted 2025-08-21; First posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Healthy Diet; Healthy Nutrition
Keywords: Healthy meal plan; Weight management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants in the intervention group will receive Green Chef meals for lunch and dinner, along with guidelines for preparing healthy breakfasts. Participants will follow this diet for 16 weeks.
  Interventions: Dietary Supplement: Green Chef Meal Delivery Program
- Control Group (No Intervention): Participants in the control group will continue their usual eating habits with no dietary changes for 16 weeks.

INTERVENTIONS:
Dietary Supplement: Green Chef Meal Delivery Program — Participants will receive Green Chef meals for lunch and dinner, delivered weekly for 16 weeks. Meals include organic produce, responsibly sourced protein, and nutritionist-approved recipes. Participants will also receive guidelines for preparing healthy breakfasts and will use smart devices to record biomarker data.
  Arms: Intervention Group

SUMMARY:
This is a 16-week, two-arm, hybrid, randomized controlled clinical trial designed to evaluate the effect of the Green Chef Calorie Smart & Brain Health meal plans on health biomarkers and perceived well-being. The study aims to measure improvements in blood lipids, body composition, weight, and blood pressure, as well as subjective health indicators through surveys.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 25 years or older.
* Participants who struggle with healthy weight management and have a desire to lose weight.
* Participants who eat takeout or at restaurants at least four times per week.
* Participants not currently using a meal kit.
* Participants who are willing to cook meals twice daily for the 16-week study period.
* Participants who are willing to cook and consume meals as instructed, fill out regular questionnaires, take regular weight and blood pressure measurements, and attend blood tests at Quest for Baseline and Endline assessments for the 16-week study period.
* Participants must not have introduced any new prescription medications, supplements, or herbal remedies targeting weight management within the past three months.
* Participants must be willing to discontinue any prescription medications, supplements, or herbal remedies that target weight management for the duration of the trial.
* Participants must agree to not introduce any new prescription medications, vitamins, minerals, nutraceuticals, or herbal supplements for the duration of the trial.
* Participants must consider themselves in good general health and not have any chronic health conditions that could impact their participation in the study.
* Participants must reside in the United States.

Exclusion Criteria:

* Individuals who have undergone surgeries or invasive treatments in the last six months or have any planned for the duration of the trial.
* Individuals who have undergone weight loss surgery.
* Individuals who have experienced dramatic weight changes (gain or loss) within the past three months.
* Individuals who consider themselves to be chronic dieters or "always on a diet" (e.g., those who have been dieting or restricting calories for a prolonged period of time or who tend to jump from one diet to the next regularly).
* Individuals with a known history of severe digestive disorders, including but not limited to acid reflux, Irritable Bowel Syndrome (IBS), Inflammatory Bowel Disease (IBD), ulcerative colitis (UC), Crohn's disease, or gastrointestinal tract surgeries.
* Individuals with a known history of any chronic illness such as hypertension, diabetes, or cancer.
* Individuals with any known allergies or hypersensitivities to foods.
* Individuals with a history of disordered eating behaviors or an eating disorder.
* Individuals who regularly take laxatives, or antacids.
* Individuals who regularly take anticoagulants (also referred to as blood thinners).
* Individuals with chronic health conditions, including oncological or psychiatric disorders, that could impact participation.
* Individuals with known serious allergic reactions requiring the use of an Epi-Pen.
* Individuals who are currently pregnant, trying to conceive, or breastfeeding.
* Individuals currently participating or planning to participate in another research study within the next 16 weeks.
* Individuals with a history of substance abuse.
* Individuals with specific dietary restrictions that make consuming the test meals impossible (e.g., pescatarian, vegetarian, vegan, Whole 30, FODMAP).
* Anyone who has taken a GLP-1 agonist in the last 3 months.

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-11-19 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Blood Lipid Biomarkers (LDL, HDL, Triglycerides) | Baseline to Week 16
  Blood lipid levels (LDL, HDL, triglycerides) will be measured at baseline and week 16 via fasting blood draws to evaluate the effect of the Green Chef meal plan on cardiovascular health.
Change in Weight and Body Composition | Baseline, Week 8, Week 16
  Body weight and composition will be measured using a Withings smart scale at baseline, week 8, and week 16 to assess changes related to the dietary intervention.
Change in Blood Pressure | Baseline, Week 8, Week 16
  Systolic and diastolic blood pressure will be measured using a Withings smart blood pressure cuff at baseline, week 8, and week 16 to assess impact of the meal plan on cardiovascular function.

SECONDARY OUTCOMES:
Change in Self-Reported Health Perceptions | Baseline, Week 4, Week 8, Week 12, Week 16
  Participants will complete surveys at 5 time points to assess subjective changes in energy, digestion, eating habits, physical appearance, and overall well-being.

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Las Vegas, Nevada, United States